CLINICAL TRIAL: NCT02942056
Title: The Effect of Cinnamon Cassia on Diabetes Control and Cardiometabolic Risk Factors in Adults With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not obtain appropriate funding or standardized manufacturing for cinnamon tablets
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Scott M. Chadderdon, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OHSU IRB # 11386
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Drug (Experimental): Randomized to cinnamon cassia 750 mg TID for 6 months. Assess HbA1c and CV risk profile
  Interventions: Drug: Cinnamon
- Placebo (Placebo Comparator): Randomized to placebo matching tablet TID for 6 months. Assess HbA1c and CV risk profile
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Cinnamon — Cinnamon tablets to treat type 2 DM
  Arms: Study Drug
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The overall goal of this proposal is to establish the efficacy of cinnamon for the treatment of T2DM. Additional aims will assess the effect of cinnamon on cardiovascular risk factors and explore novel potential mechanisms of action leading to improved insulin sensitivity. Based on previously published animal and human data we have hypothesized that six months treatment with Cinnamon cassia supplementation (2.25 grams/day) will improve glycemic control and cardio-metabolic risk factors. We believe these benefits may be mediated in part through improved insulin mediated capillary recruitment and skeletal muscle vasodilators leading to reduced insulin resistance. We will achieve our goal through completion of the following aims:

Aim 1. To demonstrate the efficacy, safety, and tolerability of oral cinnamon use (750 mg three times daily) to improve glucose control. The primary outcome will be determined as a reduction in hemglobin A1c (HbA1c) level of at least 0.5% compared to placebo.

Aim 2. To quantify effects of oral cinnamon (vs. placebo) on cardio-metabolic risk factors, including: fasting levels of plasma insulin and glucose, homeostatic model assessment of insulin resistance (HOMA-IR), lipids (total, VLDL, LDL, HDL cholesterol; triglyceride), free fatty acids, as well whole body, abdominal, and visceral adiposity as measured with dual energy x-ray absorptiometry (DEXA) imaging.

Aim 3. In this mechanistic exploratory aim, potential gastrointesitnal effects will be assessed as follows: a 3-hour oral glucose tolerance test (OGTT) with blood samples collected for insulin, glucose, C-peptide, glucagon, GLP-1, and GIP will be performed separately. Additional biochemical markers (ghrelin, PYY, pro-insulin, apo B, adinopectin) will be collected as well.

DETAILED DESCRIPTION:
Experimental Design:

This Phase 2 study will be done prospectively and will be conducted in two stages. The initial stage will be the general study and the second stage will be the sub-study. We plan to screen up to 1,000 subjects. Our enrollment goal is 250 subjects total (with 50 subjects enrolled in the sub-study and 200 subjects enrolled in the general study).

Adults will be screened from Oregon Health & Science University clinics (cardiology, internal medicine, endocrinology, obstetrics and gynecology, family practice) through Epic-based database searches and research flyer distribution. At OHSU, the Research Data Warehouse (RDW) will be used to identify potential subjects and recruitment letters will be sent out. Additional advertisement will be conducted through March Wellness and the medical exercise program. Further outreach advertising will be done through the Oregon Association of Naturopathic Physicians (OANP) website and the Naturopathic Doctor News & Reviews (NDNR) newsletter.

We will not include any vulnerable populations. We will not recruit prisoners, children, neonates, and/or adults lacking capacity.

In the event of a screen failure, the data collected in screening will be retained to avoid future re-contacting for recruitment for this study. The data will be handled in a confidential manner until destroyed at the end of enrollment.

Inclusion/Exclusion Criteria:

Recruited subjects will meet the following criteria:

Inclusion Criteria:

* Males and females ages 30-65 years of age
* Diagnosed Type 2 diabetes with a HbA1c of 6.5-9%, treated with either lifestyle alone or with metformin
* Weight stable for 3 months as defined by no greater than a 5% change.

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Use of any other diabetes treatment other than metformin within the past 3 months
* Type 1 diabetes
* HbA1c > 9% or less than< 6.5%
* Liver disease with a known diagnosis of cirrhosis
* Liver Dysfunction with AST or ALT liver enzymes > 2x upper limit of normal
* Chronic Kidney Disease with glomerular filtration rate < 45 ml/min/1.73m2
* Anemia with hematocrit < 30%
* TSH > 5 or < 0.4 mIU/L
* Coagulopathy, INR > 1.3
* Use of warfarin or other new oral anticoagulants (dabigatran, rivaroxaban, apixaban)
* Use of subcutaneous heparin, enoxaparin, dalteparin
* Use of class 1 or class 3 anti-arrhythmic medications (disopyramide, procainamide, quinidine, mexilitine, flecanide, propafenone, amiodarone, sotalol, dronedarone, dofetilide)
* Use of immunosuppressants (methotrexate, prednisone, tacrolimus, sirolimus, azathioprine, mycophenolate, cyclosporine)
* Chronic use of benzodiazepines (midazolam, alprazolam, lorezepam, temezepam, diazepam, clonazepam, chlordiazepoxide) for the past 3 months
* Chronic use of medications that may affect body weight, glucose or lipid metabolism (e.g., anti-psychotics, anti-seizure, weight loss meds) for the past 3 months
* Patients with celiac sprue or gluten sensitive individuals
* Self-report of > 3 alcoholic drinks per day
* Congestive heart failure (ejection fraction < 45%)
* Known hypersensitivity to Definity® ultrasound contrast agent (for sub-study)
* Intra-cardiac or pulmonary shunt

Screening Visit:

After receiving a verbal and graphical summary of the study, subjects may opt into the General Study or a more detailed Mechanistic Sub-Study. See below.

Baseline Visit and Week 6 to 24 Study Visits (in the General Study):

Once subjects are screened, those that have consented and are enrolled in the General Study will undergo the following tests and procedures:

1. For women of child bearing potential, a urine pregnancy test will be performed. This must be done prior to iDEXA scan, and should be done prior to randomization.
2. Complete chemistry panel for liver and kidney function, fasting insulin, complete blood count (CBC), fasting lipid panel, urine analysis, and iDEXA scan for body composition. Subject must be fasting for 8 hours. Any remaining blood samples, after being used for this study, will be stored in the repository.
3. Subjects will have an Actical monitor fit to their waist to wear for one week.
4. 24 hour food recalls will be performed by study staff. The recalls will be conducted over the phone three separate times within 14-21 days at baseline and at 24 weeks.
5. Prior to baseline visit discharge, subjects will be randomized in a double blinded fashion in a 1:1 ratio to either 750 mg of cinnamon cassia or placebo three times daily for 24 weeks.
6. Pills will be picked up and empty bottles returned for pill count by study staff at every visit.
7. After 6 weeks of treatment, subjects will have blood and urine testing for safety monitoring (liver function tests, CBC, and urine analysis).
8. After 12 weeks of treatment an HbA1c, fasting insulin, and fasting lipid panel will be drawn for an interim analysis. Repeat safety profile with a complete chemistry panel for liver and kidney function and CBC will also be obtained. Subject must be fasting for 8 hours.
9. After 24 weeks of therapy, subjects will return for a final visit in which all baseline tests and procedures will be repeated. (blood draw, urine test, iDEXA, Actical, food recalls)
10. Adverse events and concomitant medications will be reviewed.
11. Baseline visit will occur 10 ± 5 days from the screening visit
12. All follow-up visits, Weeks 6-24, will be done ± 7 days.

Baseline Visit and Week 6 to 24 Study Visits (in the Sub-Study):

Those subjects that have consented and are enrolled in the Mechanistic Sub-Study will undergo the following baseline tests and procedures:

On Day 1 of baseline testing the following tests will be performed:

1. For women of child bearing potential, a urine pregnancy test will be performed. This must be done prior to iDEXA scan, and should be done prior to randomization.
2. Complete chemistry panel for liver and kidney function, fasting insulin, CBC, fasting lipid panel, HbA1c, urine analysis, and iDEXA scan for body composition. Any remaining blood samples, after being used for this study, will be stored in the repository.

On Day 2 of baseline testing (within 1 week of Day 1) the following tests will be performed:

1. Oral glucose tolerance test with a plasma sample obtained just prior to and after glucose ingestion for GI secretory function analysis.
2. Subjects will have an Actical activity monitor fit to their waist to wear for a week.
3. 24 hour food recalls will be scheduled and performed by study staff.

Following completion of these baseline studies, subjects will be randomized in a double blinded fashion in a 1:1 ratio to either 750 mg of cinnamon cassia or placebo three times daily for 24 weeks.

At the 6 and 18 week visit the following tests will be performed: blood draw will be for safety with LFTs, CBC, and Urinalysis.

At the 12 week visit the following tests and procedures will be performed:

1. Subjects will be admitted to the CTRC for active metabolite testing.
2. Subjects will have blood testing for safety monitoring (complete chemistry panel with LFTs, CBC, and urinalysis) and an HbA1c, fasting insulin, and fasting lipid panel drawn for an interim analysis.

After 24 weeks of therapy, subjects will return for a final visit in which all baseline tests will be repeated.

Methods:

All Methods below are research related inquiries.

Dual X-Ray Absorptiometry (DEXA): Body composition (total lean and fat mass and skeletal mineral content) and body fat distribution will be measured by a trained technician in OHSU's Body Energy and Composition Core using a GE Healthcare Lunar iDEXA with encore software. Pregnancy testing will be performed in all women prior to each total body scan. If the results are positive, the participant will be withdrawn from the study and referred to her personal health care provider.

OGTT: Following an overnight fast, subjects will have an IV placed in an antecubital fossa. After at least 15 minutes of rest, three baseline samples will be obtained and the subject will then ingest 75 gm of glucose. Blood for glucose, insulin, C-peptide, glucagon, GLP-1, and GIP will be obtained at times -15, -10, -5, 0,15, 30, 60, 90, 120, and 180 minutes. Proinsulin will be measured in one of the baseline samples. Insulin sensitivity will be estimated using the Insulin Sensitivity Index (10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during OGTT]). 22 Insulin secretion capacity will be estimated using the Insulinogenic Index (insulinogenic index (delta area under the curve [AUC] insulin / delta AUC glucose). 23

Plasma Chemistries: Total lipids (total, VLDL, LDL, and HDL cholesterol; triglycerides, and apolipoprotein B) will be measured by the OHSU Lipid Lab. Complete chemistry panel, urine analysis, HbA1C, TSH, and CBC will be performed through the OHSU Core Laboratory. Insulin, glucose, C-peptide, glucagon, GLP-1, GIP, ghrelin, PYY, pro-insulin, apo B and adiponectin will be measured in the OCTRI Core Laboratory

24-Hour Diet Recall: A series of three 24-hour food recall interviews will be done by telephone by trained OCTRI Bionutrition Unit staff to determine nutrient intake. The recalls will be conducted over the phone three separate times within 14-21 days at baseline and at 6 months. The series of three calls will occur once before the beginning of the intervention phase, and again during the last week of Intervention (6 months) to ensure to the extent possible that diet habits have been maintained. The recalls will be unannounced and unscheduled so that participants are unlikely to change their normal eating habits. All interviewers will have completed a training program and met qualification standards established in the OCTRI Bionutrition Unit and based on Nutrition Data System for Research (NDSR). NDSR is a computer based software application developed at the University of Minnesota Nutrition Coordinating Center (NCC) that facilitates the collection of recalls in a standardized fashion [19]. Dietary intake data gathered by interview is governed by a multiple-pass interview approach [20]. Four distinct passes provide multiple opportunities for the participant to recall food intake. The first pass involves obtaining from the participant a listing of all foods and beverages consumed in the previous 24 hours. This listing is reviewed with the participant for completeness and correctness (second pass). The interviewer then collects detailed information about each reported food and beverage, including the amount consumed and method of preparation (third pass). Finally, the detailed information is reviewed for completeness and correctness (fourth pass).

Activity Monitors: Physical activity will be monitored using an Actical accelerometer (Mini Mitter Co., Inc., Bend, Oregon). The Actical activity monitoring device utilizes a multidirectional accelerometer to monitor the occurrence and intensity of motion. The Actical device measures 3 cm by 3 cm, weighs 17.0 grams, and is securely attached to a waistband and placed around the waist. The device can be worn and collect data for 42 days. Data are uploaded and downloaded using an ActiReader. Data include Daily Active Energy Expenditure and Total Daily Energy Expenditure. Actical's activity count data is converted into minute-by-minute energy expenditure. This is used to calculate daily caloric expenditure. Physical activity will be monitored for a seven day period at baseline, and at the 6 month time point post randomization.

Plasma Cinnamon Metabolite Identification: Plasma metabolites that constitute the active metabolite form of cinnamon will be tested while on steady state therapy at the 3 month time point. Subjects will be instructed to take their morning dose of the study drug 2 hours (+/- 30 minutes) before their scheduled study visit. They will be admitted to the clinical trial unit in the morning, if possible. Blood will be drawn for safety analysis as above as well as for active plasma metabolites. Lunch will be provided. A second blood draw for active metabolites will be obtained at 6 hours (+/- 30 minutes) after the first blood draw and just prior to the next cinnamon dose to test the difference in metabolites from 8 am to 2pm. All blood samples for active metabolites will be batched and tested at the end of the trial to maintain blinding of the study. Metabolites found to be significantly different (p<0.05) between experimental groups will be identified by searching our in-house library which contains >600 metabolites (Mass Spectrometry Metabolite Library of Standards, IROA Technologies, LLC) and >100 phytochemicals), or our LipidView database which contains >25,000 lipids. When metabolites of interest are absent from our in-house library of metabolites and the LipidView database, we will perform online database searches (METLIN; http://metlin.scripps.edu, HMDB; http://www.hmdb.ca/, and MassBank; http://www.massbank.jp/?lang=en) using their accurate masses. When available, database MS/MS spectra will be used to further confirm the identity of the metabolite. If a metabolite of interest is absent from all databases, PeakView software (AB SCIEX) will be used to create a potential list of molecular formulas matching the measured m/z value (within 15 ppm error), fragmentation pattern, and isotopic distribution (within 20% error). For many of the metabolites identified, synthetic standards can be purchased to confirm method specific MS/MS spectra, retention time, experimental m/z value, and isotopic distribution.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 30-65 years of age
* Diagnosed Type 2 diabetes with a HbA1c of 6.5-9%, treated with either lifestyle alone or with metformin
* Weight stable for 3 months as defined by no greater than a 5% change.

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Use of any other diabetes treatment other than metformin within the past 3 months
* Type 1 diabetes
* HbA1c > 9% or less than< 6.5%
* Liver disease with a known diagnosis of cirrhosis
* Liver Dysfunction with AST or ALT liver enzymes > 2x upper limit of normal
* Chronic Kidney Disease with glomerular filtration rate < 45 ml/min/1.73m2
* Anemia with hematocrit < 30%
* TSH > 5 or < 0.4 mIU/L
* Coagulopathy, INR > 1.3
* Use of warfarin or other new oral anticoagulants (dabigatran, rivaroxaban, apixaban)
* Use of subcutaneous heparin, enoxaparin, dalteparin
* Use of class 1 or class 3 anti-arrhythmic medications (disopyramide, procainamide, quinidine, mexilitine, flecanide, propafenone, amiodarone, sotalol, dronedarone, dofetilide)
* Use of immunosuppressants (methotrexate, prednisone, tacrolimus, sirolimus, azathioprine, mycophenolate, cyclosporine)
* Chronic use of benzodiazepines (midazolam, alprazolam, lorezepam, temezepam, diazepam, clonazepam, chlordiazepoxide) for the past 3 months
* Chronic use of medications that may affect body weight, glucose or lipid metabolism (e.g., anti-psychotics, anti-seizure, weight loss meds) for the past 3 months
* Patients with celiac sprue or gluten sensitive individuals
* Self-report of > 3 alcoholic drinks per day
* Congestive heart failure (ejection fraction < 45%)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Type 2 DM control | 6 months
  change in HbA1c

SECONDARY OUTCOMES:
lipid control | 6 months
  change in LDL, HDL, triglycerides
obesity | 6 months
  change in abdominal fat percentage